CLINICAL TRIAL: NCT03311984
Title: Evaluation of Anti-Xa Levels in Critically Ill Patients Receiving Low-molecular-weight Heparin for Thromboprophylaxis in China
Brief Title: Anti-Xa Levels in Critically Ill Patients Receiving Low-molecular-weight Heparin for Thromboprophylaxis in China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Chun Pan, professor, Southeast University, China
Other Study IDs: Anti-Xa Level
Record Dates: First submitted 2017-10-06; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Critically Ill; Anti-Xa
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LMWH qd: receiving Low-molecular-weight Heparin（LMWH）qd
  Interventions: Diagnostic Test: anti Xa level
- LMWH q12h: receiving Low-molecular-weight Heparin（LMWH）q12h
  Interventions: Diagnostic Test: anti Xa level

INTERVENTIONS:
Diagnostic Test: anti Xa level — monitoring the anti-Xa level according to LMWH emploing

SUMMARY:
Critically ill Patients are at high risk to develop deep venous thrombosis. However, despite receiving of a standard dose of Low-molecular-weight Heparin（LMWH）, many patients still develop life-threatening embolism. The purpose of this study is to evaluate the anti-Xa levels of different dosing regimens of LMWH in critically ill patients in China.

ELIGIBILITY:
Inclusion Criteria:

* Adult Critically ill patients

Exclusion Criteria:

* Contraindication to use of LMWH. Intracranial bleeding/stroke, hematoma or bleeding disorder. Use Heparin anticoagulant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Critically ill patients Receiving Low-molecular-weight Heparin for Thromboprophylaxis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-05-30 (Estimated)

PRIMARY OUTCOMES:
Anti-Xa Levels | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Changde Wu, Nanjing, Jiangsu, China